CLINICAL TRIAL: NCT05356351
Title: An Open-label, Single-arm, Multicenter Phase II Clinical Study： Evaluating RC48-ADC Combined With Triplizumab in the Neoadjuvant Treatment of Her2-positive Muscle-invasive Bladder Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Xiangya Hospital of Central South University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Southwest Hospital, China (Other); Tongji Hospital (Other); Chongqing University Cancer Hospital (Other); Hunan Cancer Hospital (Other); The First Affiliated Hospital of Air Force Medicial University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-TA001
Record Dates: First submitted 2022-04-18; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-02

CONDITIONS: Neoadjuvant Treatment of Her2-positive Muscle-invasive Bladder Cance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- test group (Experimental): RC48-ADC 2.0 mg/kg）D1,Triplizumab 3mg/kg D2，Q2W
  Interventions: Drug: RC48- ADC

INTERVENTIONS:
Drug: RC48- ADC — RC48-ADC 2.0 mg/kg D1,Triplizumab 3mg/kg D2，Q2W
  Other Names: Triplizumab

SUMMARY:
An Open-label, Single-arm, Multicenter Phase II Clinical Study： Evaluating RC48-ADC Combined With Triplizumab in the Neoadjuvant Treatment of Her2-positive Muscle-invasive Bladder Cancer.It's arm to evaluate the neoadjuvant treatment of Her2-positive Muscle-invasive Bladder Cancer in patients with objective response rate (ORR),Duration of response (DoR) , progression-free survival (PFS), overall survival (OS), and safety.

DETAILED DESCRIPTION:
Objective response rate (ORR), Duration of response (DoR) (according to RECIST 1.1 Standard Edition)，progression-free survival (PFS), overall survival (OS), quality of life (QoL)and safety. Evaluation once every 2 weeks before cystectomy, If the efficacy results of the evaluation are complete response (CR) or partial response (PR), confirmed imaging efficacy at 9 weeks after the initial assessment ， efficacy evaluation time window of ± 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is volunteer to participate, and the subject must signed an informed consent form (ICF), indicating that it understands the purpose of this study and the required procedures, and is willing to participate in the study. Subjects must be willing and abide by prohibition and restrictions specified in the research program; Subjects are willing and able to follow the trial and follow-up procedures
2. Patients with invasive bladder cancer are prepared for radical cystectomy (standard lymph node dissection);
3. Age ≥ 18 years old and ≤ 75 years old;
4. Clinical stage T2-T4aN0M0 (assessed by CT/MR/PET-CT);
5. Pathological was confirmed urothelial carcinoma by TURBT, HER2 overexpression confirmed by pathological biopsy: IHC2+ or IHC3+(central laboratory verification) andthe physical condition was not suitable for neoadjuvant chemotherapy ( pathological permit urothelial carcinoma Combined with other variant subtypes, with urothelial carcinoma as the main type) or refused neoadjuvant chemotherapy;
6. ECOG score ≤ 1;
7. After TURBT, residual tumor (measurable according to RECIST 1.1 criteria) is present;
8. The important laboratory examination indexes meet the following requirements:

   1. Hemoglobin ≥ 90g/L.
   2. Absolute neutrophil count (ANC) ≥ 1.5 × 109 / L.
   3. Platelet ≥ 100 × 109 / L.
   4. 3.5mmol/L ≤ serum potassium ≤ 5.5mmol/L.
   5. Liver function index: ALT, AST ≤ 1.5 times the upper limit of normal value (ULN), TBIL ≤ 1.5ULN.
   6. Subjects with Serum creatinine≤ 1.5× ULN
   7. The left ventricular ejection fraction (LVEF) was 50%.
9. Female subjects should be surgically sterilized or postmenopausal, or agree to use at least one medically approved contraceptive method (such as intrauterine device, contraceptive or condom) during the study treatment and within 6 months after the end of the study treatment period. The blood pregnancy test must be negative within 7 days before the study, and it must be non-lactation. Male subjects should agree to use at least one medically approved contraceptive method (such as condoms, abstinence, etc.) during the study treatment period and within 6 months after the end of the study treatment period.

Exclusion Criteria:

1. Had received live attenuated vaccine or had serious infection or planned to receive any vaccine during the study period4 weeks before entering the group.
2. Received antineoplastic therapy within 6 months before the start of the study, including chemotherapy, radiotherapy, targeted therapy, immunotherapy and clinical research antineoplastic drug therapy.
3. Uncontrollable concomitant diseases, including, but not limited to, persistent infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, arrhythmia, interstitial lung disease, severe chronic gastrointestinal disease associated with diarrhoea, or mental illness / social conditions, which will limit compliance with research requirements, significantly increase the risk of AE or impair the patient's ability to write informed consent.The results of HIVAb test were positive;with active bleeding or new thrombotic disease who are taking therapeutic anticoagulants or who have a tendency to bleed
4. Patients with RC48-ADC /PD-1 allergy or hypersensitivity, patients with autoimmune diseases;
5. HBsAg or HBcAb test results are positive, while HBVDNA copies are positive; HCVAb test results are positive (only if the PCR test result of HCVRNA is negative);Systemic corticosteroids or other systemic immunosuppressive drugs are used before enrollment, or systemic immunosuppressive drugs are expected to be needed during the trial;
6. Serious arteriovenous thrombosis or cardio-cerebrovascular accidents occurred within 1 year before administration, such as deep venous thrombosis, pulmonary embolism, cerebral infarction, cerebral hemorrhage, myocardial infarction, etc., except for lacunar infarction that is asymptomatic and does not require clinical intervention;with active bleeding or new thrombotic disease who are taking therapeutic anticoagulants or who have a tendency to bleed.
7. Active/known/suspected autoimmune disease, history of primary immunodeficiency,Previous allogeneic hematopoietic stem cell transplantation;
8. Diagnosed with other malignancies within 5 years
9. Pregnant or lactating women.
10. Patients with missing main observation indicators, incomplete research data, incomplete follow-up data or failure to follow the research protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Pathological response (PaR) rate | Up to approximately 6 months
  Pathological response (PaR) rate per central pathology review
recommended dose for phase II safety (RP2D) | Up to approximately 6 months
  tolerability
Incidence of adverse events and serious adverse events | Up to approximately 6 months
  safety

SECONDARY OUTCOMES:
The pathological complete response | Up to approximately 6 months
  The pathological complete response rate refers to all target lesions disappear
Progression free survival | Up to approximately 24 months
  Follow-up was made after the first month after the operation, and then with an every three months until the tumor relapsed or progress
Overall survival | Up to approximately 48 months
  The time from start of study treatment to date of death due to any cause
Duration of response | Up to approximately 24 months
  This is the time from when the tumor begins to respond to treatment until the disease gets worse

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol